CLINICAL TRIAL: NCT00911508
Title: Catheter Ablation vs Anti-arrhythmic Drug Therapy for Atrial Fibrillation Trial
Acronym: CABANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Abbott Medical Devices (Industry); Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Douglas L. Packer, MD, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-004616; U01HL089709 (NIH)
Record Dates: First submitted 2009-05-28; First posted 2009-06-02 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Atrial Fibrillation; Left Atrial Ablation; Pulmonary Vein Isolation; Catheter Ablation; Antiarrhythmic Drug Therapy
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left Atrial Ablation (Active Comparator): Pulmonary vein isolation using a circumferential ablative approach in the left atrium. Ablation may be performed using circular mapping catheter-guided ablation, antral isolation using a circular guided approach, or wide area circumferential ablation.
  Interventions: Device: Left atrial ablation
- Rate or Rhythm Control Therapy (Active Comparator): Current state-of-the-art drug therapy for atrial fibrillation (rate control or rhythm control). Treating physicians will be encouraged to follow the American College of Cardiology / American Heart Association / European Society of Cardiology Atrial Fibrillation Guidelines with regard to drug therapy for atrial fibrillation. The specific choice of rate control versus rhythm control drug therapy and the specific drugs to be used will ultimately be left to the discretion of the treating physician.
  Interventions: Drug: Rate or Rhythm Control Therapy

INTERVENTIONS:
Device: Left atrial ablation — St. Jude: Livewire TC™ , Therapy™ Dual / Thermocouple, Safire,Therapy Cool Path
  Biosense Webster: NAVI-STAR, NAVI-STAR/NAVI-STAR DS, Celsius Braided/Long Tip, NAVI-STAR™ and Celsius™ ThermoCool, NAVI-STAR® RMT, Celsius® RMT, ThermoCool® SF
  Medtronic CryoCath LP: Freezor®/Freezor MAX®, Artic Front®, Cardiac Ablation System
  Bard: Stinger
  Boston Scientific: Blazer II RF/XP, Blazer RPM, Chilli II Cooled, SteeroCath
  Arms: Left Atrial Ablation
Drug: Rate or Rhythm Control Therapy — Rate control: Metoprolol 50-100mg, Atenolol 50-100mg, Propranolol 40-80mg, Acebutolol 200-300mg, Carvedilol 6.25-25mg, Diltiazem 180-240mg, Verapamil 180-240mg, Digoxin 0.125-0.25mg
  Rhythm control: Propafenone 450-625mg, Flecainide 200-300mg, Sotalol 240-320mg, Dofetilide 500-1000mcg, Amiodarone 200-400mg, Quinidine 600-900mg, Dronedarone 800mg
  Arms: Rate or Rhythm Control Therapy

SUMMARY:
The (Catheter Ablation Versus Anti-arrhythmic Drug Therapy for Atrial Fibrillation Trial) CABANA Trial has the overall goal of establishing the appropriate roles for medical and ablative intervention for atrial fibrillation (AF). The CABANA Trial is designed to test the hypothesis that the treatment strategy of left atrial catheter ablation for the purpose of eliminating atrial fibrillation (AF) will be superior to current state-of-the-art therapy with either rate control or rhythm control drugs for decreasing the incidence of the composite endpoint of total mortality, disabling stroke, serious bleeding, or cardiac arrest in patients with untreated or incompletely treated AF.

DETAILED DESCRIPTION:
The need for this trial arises out of 1) the rapidly increasing number of pts > 60 years of age with AF accompanied by symptoms and morbidity, 2) the failure of anti-arrhythmic drug therapy to maintain sinus rhythm and reduce mortality, 3) the rapidly increasing application of radio-frequency catheter ablation without appropriate evidence-based validation, and 4) the expanding impact of AF on health care costs.

This study will randomize up to 2200 patients to a strategy of catheter ablation versus pharmacologic therapy with rate or rhythm control drugs. Each pt will have 1) characteristics similar to AFFIRM pts (≥65 yo or <65 with >1 risk factor for stroke, 2) Documented AF warranting treatment, and 3) Eligibility for both catheter ablation and ≥2 anti-arrhythmic or ≥2 rate control drugs. Pts will be followed every 6 months for an average of approximately 5 years and will undergo repeat trans-telephonic monitor, Holter monitor, and CT/MR studies to assess the impact of treatment.

The CABANA trial will disclose the role of medical and non-pharmacologic therapies for AF, establish the cost and impact of therapy on quality of life and will help determine if AF is a modifiable risk factor for increased mortality.

ELIGIBILITY:
Inclusion Criteria:

* Over the preceding 6 months have:

  1. ≥2 paroxysmal (electrocardiographic documentation of at least 1) atrial fibrillation (AF) episodes lasting ≥1 hour in duration: (that terminate spontaneously within 7 days or cardioversion is performed within 48h of AF onset): or
  2. electrocardiographic documentation of 1 persistent AF episode: (sustained for ≥7 days or cardioversion is performed more than 48h after AF onset): or
  3. electrocardiographic documentation of 1 longstanding persistent AF episode: (continuous AF of duration >1 year).
* Warrant active therapy (within the past 3 months) beyond simple ongoing observation
* Be eligible for catheter ablation and ≥2 sequential rhythm control and/or ≥2 rate control drugs.
* Be ≥65 yrs of age, or <65 yrs with one or more of the following risk factors for stroke: Hypertension (treated and/or defined as a blood pressure >140/90 mmHg) [90], Diabetes (treated and/or defined as a fasting glucose ≥126 mg/dl) [91], Congestive heart failure (including systolic or diastolic heart failure), Prior stroke, transient ischemic attack or systemic emboli, Atherosclerotic vascular disease (previous myocardial infarction (MI), peripheral arterial disease or aortic plaque), left atrial (LA) size >5.0 cm (or volume index ≥40 cc/m2), or ejection fraction (EF) ≤35.
* Have the capacity to understand and sign an informed consent form.
* Be ≥18 years of age.

  * NOTE- Subjects <65 yrs of age whose only risk factor is hypertension must have a second risk factor or left ventricular (LV) hypertrophy to qualify.Patients receiving new drug therapy initiated within the previous 3 months may continue that therapy if randomized to the drug therapy arm. Patients may have documented atrial flutter in addition to atrial fibrillation and remain eligible for enrollment.

Exclusion Criteria:

* Lone AF in the absence of risk factors for stroke in patients <65 years of age
* Patients who in the opinion of the managing clinician should not yet receive any therapy for AF
* Patients who have failed >2 membrane active anti-arrhythmic drugs at a therapeutic dose due to inefficacy or side effects (Table 5.2.2)
* An efficacy failure of full dose amiodarone treatment >8 weeks duration at any time
* Reversible causes of AF including thyroid disorders, acute alcohol intoxication, recent major surgical procedures, or trauma
* Recent cardiac events including MI, percutaneous intervention (PCI), or valve or bypass surgery in the preceding 3 months
* Hypertrophic obstructive cardiomyopathy (outflow track)
* Class IV angina or Class IV congestive heart failure (CHF) (including past or planned heart transplantation)
* Other arrhythmias mandating anti-arrhythmic drug therapy (i.e. ventricular tachycardia (VT), ventricular fibrillation (VF))
* Heritable arrhythmias or increased risk for torsade de pointes with class I or III drugs
* Prior LA catheter ablation with the intention of treating AF
* Prior surgical interventions for AF such as the MAZE procedure
* Prior AV nodal ablation
* Patients with other arrhythmias requiring ablative therapy
* Contraindication to appropriate anti-coagulation therapy
* Renal failure requiring dialysis
* Medical conditions limiting expected survival to <1 year
* Women of childbearing potential (unless post-menopausal or surgically sterile)
* Participation in any other clinical mortality trial (Participation in other non-mortality trials should be reviewed with the clinical trial management center)
* Unable to give informed consent

  * NOTE- Prior ablation of the cavo-tricuspid isthmus alone is not an exclusion if the patient develops subsequent recurrent AF. Planned atrial flutter ablation in combination with the left atrial ablation is not an exclusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2204 (Actual)
Dates: Start 2009-11-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas L. Packer, M.D., Principal Investigator — Mayo Clinic; Kerry L. Lee, Ph.D., Principal Investigator — Duke Clinical Research Institute; Daniel B. Mark, M.D., MPH, Principal Investigator — Duke Clinical Research Institute; Rich A. Robb, Ph.D. Phy, Principal Investigator — Mayo Clinic; Yves D. Rosenberg, M.D., MPH, Study Chair — National Heart, Lung, and Blood Institute (NHLBI)
Locations (118):
- United States (76):
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Good Samaritan Hospital, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California at San Francisco Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Penrose Saint Francis Health Services, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Miami Hospital, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Northside Hospital and Heart Institute, St. Petersburg, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Florida Heart Rhythm-University of South Florida College of Medicine, Tampa, Florida
  - Georgia Regents University, Augusta, Georgia
  - Georgia Arrhythmia Consultants & Research Institute, Macon, Georgia
  - Alexian Brothers Medical Center, Barrington, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Mercy Medical Center-Iowa Heart Center, West Des Moines, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Joseph Mercy Hospital, Ypsilanti, Michigan
  - Minneapolis V.A. Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Park Nicollet Methodist Hospital, Saint Louis Park, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - Saint John's Mercy Heart Health Center, St Louis, Missouri
  - Saint Louis Heart and Vascular, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Associates in Cardiology, Albany, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Stony Brook University Hospital and Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Sanger Clinic, PA, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Geisinger Wyoming Valley Medical Center, Danville, Pennsylvania
  - Penn State University Cardiovascular Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - V.A. Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Greenville Hospital System University Medical Center, Greenville, South Carolina
  - Memorial Health Care System, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - University of Texas Health Science Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Intermountain Medical Center-LDS Hospital, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Hospital Center - Arlington, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Swedish Medical Center - Providence Campus, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cardiac Study Center, Tacoma, Washington
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - University of Western Ontario - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
- China (5):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Beijing Anzhen Hospital, Beijing
  - Fuwai Hospital, Beijing
- Czechia (4):
  - Na Homolce Hospital, Prague, Prague
  - Saint Anne's University Hospital, ICRC, Brno
  - Charles University, Prague
  - Clinic of Cardiology IKEM Medical Institute, Prague
- Germany (14):
  - University Hospital of Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum Coburg, Coburg, Bavaria
  - Universitares Herrzentrum Hamburg, Hamburg, Freie-Hansestadt Hamburg
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Technische Universitat Dresden, Dresden, Saxony
  - Kerckhoff Klinik, Bad Nauheim
  - Praxisklinik Herz and GefaBe, Dresden
  - CCB - Cardioaniologisches Centrum Bethanien, Frankfurt
  - Georg-August-University, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Saint Vincentius-Kliniken, Karlsruhe
  - Herzzentrum Leipzig, Leipzig
  - Universitat Rostock, Rostock
- Italy (3):
  - Policlinico San Donato Center of Clinical Arrhythmia and Electrophysiology, San Donato Milanese, Lombardy
  - Policlinico Multimedical Cardiology and Arrhythmia Centre, Milan
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Russia (4):
  - Research Institute of Circulation of Pathology, Novosibirsk, Novosibirsk Oblast
  - Clinical Hospital # 83 under the Federal Medical and Biological Agency, Moscow
  - Bakoulev Scientific Center for Cardiovascular Surgery, Moscow
  - Scientific Research Institute of Cardiology of Ministry of Health of Russian Foundation, Tomsk
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
- United Kingdom (4):
  - Golden Jubilee Hospital, Glasgow
  - Saint Bartholomew's Hospital, London
  - Saint George's Hospital Medical School, London
  - Saint Mary's Hospital, London

REFERENCES:
- [Derived] Zhao M, Chen Y, Li M, Jiang C, Wang Z, Liu H, He L, Sang C, Du X, Dong J, Packer DL, Ma C, Lip GYH. Impact of diagnosis to ablation time on clinical outcomes in patients with atrial fibrillation: post hoc analysis of the CABANA trial. BMC Med. 2026 Jan 12. doi: 10.1186/s12916-026-04615-3. Online ahead of print. PMID 41526927
- [Derived] Wu Q, Wang L, Li Y, Liang Z, Li Q, Liu X, Yin Y, Liu Y, Hu Z, Gao H, Zhang T, Wang Y. Prognostic impact of mitral regurgitation in elderly patients with atrial fibrillation: results from the CABANA trial. Open Heart. 2025 Nov 27;12(2):e003478. doi: 10.1136/openhrt-2025-003478. PMID 41314687
- [Derived] Chen Y, Soler-Espejo E, Zhao M, Li W, Liu H, Gue Y, McDowell G, Packer DL, Lip GYH. Association between comorbidity burden and outcomes of catheter ablation vs. medical therapy for atrial fibrillation: insights from the CABANA trial. Europace. 2025 Dec 1;27(12):euaf292. doi: 10.1093/europace/euaf292. PMID 41213867
- [Derived] Wang Z, Wu Y, Jiang C, He L, Zhou N, Sang C, Dong J, Ma C. Catheter Ablation vs Drug Therapy in Patients With Atrial Fibrillation and Nonmodifiable Recurrence Risk Factors: A Secondary Analysis of the CABANA Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528124. doi: 10.1001/jamanetworkopen.2025.28124. PMID 40839264
- [Derived] Zhang J, Wang L, Li Y, Li Q, Liu X, Weng S, Yin Y, Liang Z, Zhang T, Wang Y. Atrial fibrillation phenotypes identified through cluster analysis in the CABANA study. Int J Cardiol. 2025 Nov 1;438:133606. doi: 10.1016/j.ijcard.2025.133606. Epub 2025 Jul 9. PMID 40645418
- [Derived] Martens P, Augusto SN Jr, Erzeel J, Pison L, Mullens W, Tang WHW. Effects of Atrial Fibrillation Ablation for Heart Failure With Preserved Ejection Fraction: Insights From CABANA. JACC Heart Fail. 2025 May;13(5):785-794. doi: 10.1016/j.jchf.2025.01.029. Epub 2025 Apr 16. PMID 40243977
- [Derived] Bunch TJ, Poole JE, Silverstein AP, Lee KL, Al-Khalidi HR, Hindricks G, Romanov A, Pokushalov E, Bahnson TD, Daniels MR, Piccini JP, Mark DB, Packer DL; CABANA Investigators. Prognostic Impact of Sinus Rhythm in Atrial Fibrillation Patients: Separating Rhythm Outcomes From Randomized Strategy Findings From the CABANA Trial. Circ Arrhythm Electrophysiol. 2024 May;17(5):e012697. doi: 10.1161/CIRCEP.123.012697. Epub 2024 Apr 17. PMID 38629286
- [Derived] Cappato R, Mark DB, Silverstein AP, Noseworthy PA, Bonitta G, Poole JE, Piccini JP, Bahnson TD, Daniels MR, Al-Khalidi HR, Lee KL, Packer DL; CABANA Investigators. Regional differences in outcomes with ablation versus drug therapy for atrial fibrillation: Results from the CABANA trial. Am Heart J. 2024 Apr;270:103-116. doi: 10.1016/j.ahj.2024.01.009. Epub 2024 Feb 1. PMID 38307365
- [Derived] Zeitler EP, Li Y, Silverstein AP, Russo AM, Poole JE, Daniels MR, Al-Khalidi HR, Lee KL, Bahnson TD, Anstrom KJ, Packer DL, Mark DB; CABANA Investigators. Effects of Ablation Versus Drug Therapy on Quality of Life by Sex in Atrial Fibrillation: Results From the CABANA Trial. J Am Heart Assoc. 2023 Feb 7;12(3):e027871. doi: 10.1161/JAHA.122.027871. Epub 2023 Jan 23. PMID 36688367
- [Derived] Monahan KH, Bunch TJ, Mark DB, Poole JE, Bahnson TD, Al-Khalidi HR, Silverstein AP, Daniels MR, Lee KL, Packer DL; CABANA Investigators. Influence of atrial fibrillation type on outcomes of ablation vs. drug therapy: results from CABANA. Europace. 2022 Oct 13;24(9):1430-1440. doi: 10.1093/europace/euac055. PMID 35640922
- [Derived] Bahnson TD, Giczewska A, Mark DB, Russo AM, Monahan KH, Al-Khalidi HR, Silverstein AP, Poole JE, Lee KL, Packer DL; CABANA Investigators. Association Between Age and Outcomes of Catheter Ablation Versus Medical Therapy for Atrial Fibrillation: Results From the CABANA Trial. Circulation. 2022 Mar 15;145(11):796-804. doi: 10.1161/CIRCULATIONAHA.121.055297. Epub 2021 Dec 22. PMID 34933570
- [Derived] Thomas KL, Al-Khalidi HR, Silverstein AP, Monahan KH, Bahnson TD, Poole JE, Mark DB, Packer DL; CABANA Investigators. Ablation Versus Drug Therapy for Atrial Fibrillation in Racial and Ethnic Minorities. J Am Coll Cardiol. 2021 Jul 13;78(2):126-138. doi: 10.1016/j.jacc.2021.04.092. PMID 34238436
- [Derived] Rettmann ME, Holmes DR 3rd, Monahan KH, Breen JF, Bahnson TD, Mark DB, Poole JE, Ellis AM, Silverstein AP, Al-Khalidi HR, Lee KL, Robb RA, Packer DL; CABANA Imaging Investigators. Treatment-Related Changes in Left Atrial Structure in Atrial Fibrillation: Findings From the CABANA Imaging Substudy. Circ Arrhythm Electrophysiol. 2021 May;14(5):e008540. doi: 10.1161/CIRCEP.120.008540. Epub 2021 Apr 13. PMID 33848199
- [Derived] Packer DL, Piccini JP, Monahan KH, Al-Khalidi HR, Silverstein AP, Noseworthy PA, Poole JE, Bahnson TD, Lee KL, Mark DB; CABANA Investigators. Ablation Versus Drug Therapy for Atrial Fibrillation in Heart Failure: Results From the CABANA Trial. Circulation. 2021 Apr 6;143(14):1377-1390. doi: 10.1161/CIRCULATIONAHA.120.050991. Epub 2021 Feb 8. PMID 33554614
- [Derived] Russo AM, Zeitler EP, Giczewska A, Silverstein AP, Al-Khalidi HR, Cha YM, Monahan KH, Bahnson TD, Mark DB, Packer DL, Poole JE; CABANA Investigators. Association Between Sex and Treatment Outcomes of Atrial Fibrillation Ablation Versus Drug Therapy: Results From the CABANA Trial. Circulation. 2021 Feb 16;143(7):661-672. doi: 10.1161/CIRCULATIONAHA.120.051558. Epub 2021 Jan 27. PMID 33499668
- [Derived] Poole JE, Bahnson TD, Monahan KH, Johnson G, Rostami H, Silverstein AP, Al-Khalidi HR, Rosenberg Y, Mark DB, Lee KL, Packer DL; CABANA Investigators and ECG Rhythm Core Lab. Recurrence of Atrial Fibrillation After Catheter Ablation or Antiarrhythmic Drug Therapy in the CABANA Trial. J Am Coll Cardiol. 2020 Jun 30;75(25):3105-3118. doi: 10.1016/j.jacc.2020.04.065. PMID 32586583
- [Derived] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766
- [Derived] Mark DB, Anstrom KJ, Sheng S, Piccini JP, Baloch KN, Monahan KH, Daniels MR, Bahnson TD, Poole JE, Rosenberg Y, Lee KL, Packer DL; CABANA Investigators. Effect of Catheter Ablation vs Medical Therapy on Quality of Life Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1275-1285. doi: 10.1001/jama.2019.0692. PMID 30874716
- [Derived] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Moretz K, Poole JE, Mascette A, Rosenberg Y, Jeffries N, Al-Khalidi HR, Lee KL; CABANA Investigators. Catheter Ablation versus Antiarrhythmic Drug Therapy for Atrial Fibrillation (CABANA) Trial: Study Rationale and Design. Am Heart J. 2018 May;199:192-199. doi: 10.1016/j.ahj.2018.02.015. Epub 2018 Mar 7. PMID 29754661
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2009 and April 2016, 2204, patients with atrial fibrillation from 126 sites across 10 countries, were randomized in equal proportions to either catheter ablation or drug therapy, using permuted block randomization with stratification by clinical site.
Groups:
- Left Atrial Ablation: All patients randomized to the ablation group were required to undergo left atrial pulmonary vein isolation. The addition of ancillary ablation techniques including linear, ganglion plexus, and electrogram-based approaches were left to the discretion of the investigators.
- Rate or Rhythm Control Therapy: All patients randomized to drug therapy, were treated with standard rhythm and/or rate control drugs selected in accordance with contemporary guidelines, according to investigator discretion.
Period: Overall Study
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Started | 1108 | 1096
Completed | 1002 | 966
Not Completed | 106 | 130
Not completed — Lost to Follow-up | 27 | 18
Not completed — Withdrawal by Subject | 79 | 112

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy | Total
Number analyzed (Participants) | 1108 | 1096 | 2204
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age | 68 [62 to 72] | 67 [62 to 72] | 68 [62 to 72]
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 375 | 391 | 766
  65 to <75 years old | 577 | 553 | 1130
  ≥ 75 years old | 156 | 152 | 308
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413 | 406 | 819
  Male | 695 | 690 | 1385
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 42 | 42 | 84
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 39 | 38 | 77
  White | 1018 | 1007 | 2025
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 28 | 24 | 52
  South Korea | 8 | 10 | 18
  United States | 625 | 608 | 1233
  Czechia | 18 | 23 | 41
  China | 21 | 22 | 43
  Italy | 27 | 27 | 54
  United Kingdom | 21 | 18 | 39
  Australia | 7 | 6 | 13
  Germany | 216 | 219 | 435
  Russia | 137 | 139 | 276
Atrial fibrillation type at time of enrollment [Count of Participants; unit: Participants] — Type of AF (paroxysmal = AF episodes lasting ≥1 hour in duration that terminates spontaneously within 7 days or cardioversion is performed within 48h of AF onset; Persistent = AF episode sustained for ≥7 days or cardioversion is performed more than 48h after AF onset; Longstanding Persistent = continuous AF of duration >1 year. Population: One patient randomized to Rate or Rhythm Control Therapy withdrew consent on the same day that signed consent was obtained. No baseline or additional data was recorded.
  Participants
    number analyzed (Participants) | 1108 | 1095 | 2203
    Paroxysmal | 470 | 476 | 946
    Persistent | 524 | 518 | 1042
    Long-standing persistent | 114 | 101 | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Total Mortality, Disabling Stroke, Serious Bleeding, or Cardiac Arrest in Patients Warranting Therapy for AF.
Description: All events for each component of the primary endpoint were reviewed and adjudicated in a blinded fashion by an independent clinical events committee using prospectively determined event definitions. Death was defined as all-cause mortality, disabling stroke (including intracranial bleeding) as an irreversible physical limitation defined by a Rankin Stroke Scale ≥2, and serious bleeding as bleeding accompanied by hemodynamic compromise that required surgical intervention or a transfusion of ≥3 units of blood.
Time Frame: From date of enrollment until time-to-first event over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 89 | 101
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.65 to 1.15]

2. Secondary Outcome: Number of Participants With All-cause Mortality
Description: All deaths were reviewed and adjudicated by the Clinical Events Committee
Time Frame: From date of enrollment until date of death over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 58 | 67
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.60 to 1.21]

3. Secondary Outcome: Number of Participants With Mortality or Cardiovascular (CV) Hospitalization
Description: Hospitalization was characterized by the site principal investigator (PI) and reported as part of the hospitalization case report form.
Time Frame: From date of enrollment until time-to-first event of death or CV hospitalization over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 573 | 637
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.74 to 0.93]

4. Secondary Outcome: Number of Participants With Mortality, Disabling Stroke, or CV Hospitalization (for Heart Failure or Acute Ischemic Events)
Description: Disabling stroke (including intracranial bleeding) was defined as an irreversible physical limitation defined by a Rankin Stroke Scale ≥2 and the reason for hospitalization was characterized by the site PI and reported as part of the hospitalization case report form.
Time Frame: From date of enrollment until time-to-first event of death, stroke, or CV hospitalization (for heart failure or acute ischemic event) over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 170 | 189
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.72 to 1.09]

5. Secondary Outcome: Number of Participants With Cardiovascular Death
Description: Cardiovascular death as determined by the Clinical Events Committee based on the available data provided by the Principal Investigator
Time Frame: From date of enrollment until date of a cardiovascular death over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 22 | 23
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.94, 95% CI 2-sided [0.53 to 1.68]

6. Secondary Outcome: Number of Participants With Cardiovascular Death or Disabling Stroke
Description: Disabling stroke (including intracranial bleeding) was defined as an irreversible physical limitation defined by a Rankin Stroke Scale ≥2.
Time Frame: From date of enrollment until time-to-first event of a cardiovascular death or disabling stroke over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 24 | 27
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.51 to 1.51]

7. Secondary Outcome: Number of Participants With an Arrhythmic Death or Cardiac Arrest
Description: All deaths and cardiac arrest events were adjudicated by the Clinical Events Committee
Time Frame: From date of enrollment until time-to-first event for an arrhythmic death or cardiac arrest over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 10 | 13
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.76, 95% CI 2-sided [0.33 to 1.72]

8. Secondary Outcome: Number of Participants With Heart Failure Death
Description: All deaths were categorized and adjudicated by the Clinical Events Committee
Time Frame: From date of enrollment until date of heart failure death over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 8 | 7
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.41 to 3.09]

9. Secondary Outcome: Number of Participants Free From Recurrent Atrial Fibrillation (AF) Following the 90 Day Blanking Period
Description: Data from patients using the study provided ECG event recording system were analyzed. A 30-second episode of AF in either group, confirmed through blinded review by an ECG Core Lab Committee was used for defining the endpoint of recurrent AF.
Time Frame: From date of therapy initiation until date of first AF recurrence following a 90 day wait (blanking) period over a median follow-up of 48.5 months.
Population: Subjects were analyzed in the post-blanking period if randomized treatment occurred and the subject did not die, withdraw, or get lost to follow-up before the end of the 90 day blanking period.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 611 | 629
Participants | 305 | 437
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.52, 95% CI 2-sided [0.45 to 0.60]

10. Secondary Outcome: Number of Participants With Cardiovascular Hospitalization
Description: The reason for hospitalization was characterized by the site PI and reported as part of the hospitalization case report form.
Time Frame: From date of enrollment until date of cardiovascular hospitalization over a median follow-up of 48.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1108 | 1096
Participants | 556 | 605
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; Test type: Superiority; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.77 to 0.97]

11. Secondary Outcome: Changes in Quality of Life Measures - AFEQT
Description: Atrial Fibrillation Effect on Quality of Life (AFEQT) Overall Score (Scale: 0 = complete disability, 100 = no disability). The AFEQT is a 21-item AF-specific, health-related QOL questionnaire designed to assess the effect of atrial fibrillation on patient quality of life. The AFEQT has an Overall Score (calculated from 18 of the questions) and subscale scores in three domains: symptoms, daily activities, and treatment concern. Overall and subscale scores range from 0 (corresponds to complete disability) to 100 (no AF-related disability).
Time Frame: Baseline ,12 month, 5 years
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1084 | 1078
units on a scale
  Baseline | 62.9 (20.5) | 63.1 (20.6)
  12 Month: number analyzed (Participants) | 915 | 903
  12 Month | 86.4 (16.5) | 80.9 (18.5)
  5 Year: number analyzed (Participants) | 329 | 320
  5 Year | 86.2 (16.2) | 83.3 (18.6)
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 12 Month; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 5.3, 95% CI 2-sided [3.7 to 6.9]
Statistical Analysis 2: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 5 Years; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 3.4, 95% CI 2-sided [2.1 to 4.8]

12. Secondary Outcome: Changes in Quality of Life Measures - MAFSI Frequency Score
Description: The Mayo AF-Specific Symptom Inventory (MAFSI) is a questionnaire comprised of a 10-item AF symptom checklist that asked about both the frequency and severity of each symptom. MAFSI frequency of symptoms over the past month was recorded as 0 (never), 1 (rarely), 2 (sometimes), 3 (often), and 4 (always) for each of the 10 items listed in the questionnaire. The 10 item responses were summed for a total Frequency Score that ranged from 0 (no AF symptoms) to 40 (worst score).
Time Frame: Baseline, 12 Month, 5 Year
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1069 | 1061
units on a scale
  Baseline | 11.8 (6.2) | 11.9 (6.4)
  12 Month: number analyzed (Participants) | 828 | 831
  12 Month | 6.4 (6.0) | 8.1 (6.3)
  5 Year: number analyzed (Participants) | 279 | 295
  5 Year | 5.8 (5.7) | 7.0 (6.3)
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 12 Month; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.3 to -1.2]
Statistical Analysis 2: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 5 Year; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.4, 95% CI 2-sided [-1.9 to -0.9]

13. Secondary Outcome: Changes in Quality of Life Measures - MAFSI Severity Score
Description: The Mayo AF-Specific Symptom Inventory (MAFSI) is a questionnaire comprised of a 10-item AF symptom checklist that asked about both the frequency and severity of each symptom. MAFSI severity scores over the past month were recorded as 1 (mild), 2 (moderate), and 3 (extreme) for each of the 10 items listed in the questionnaire. The 10 items items were then summed for the total Severity Score that ranged from 0 (no AF symptoms) to 30 (most severe AF symptoms).
Time Frame: Baseline, 12 Month, 5 Year
Population: Only patients with questionnaire data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1066 | 1056
units on a scale
  Baseline | 9.3 (4.9) | 9.3 (5.1)
  12 Month: number analyzed (Participants) | 827 | 830
  12 Month | 5.0 (4.7) | 6.5 (5.1)
  5 year: number analyzed (Participants) | 279 | 295
  5 year | 4.6 (4.7) | 5.6 (4.9)
Statistical Analysis 1: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 12 Month; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.0 to -1.1]
Statistical Analysis 2: Comparison: Left Atrial Ablation vs Rate or Rhythm Control Therapy; 5 Year; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.7 to -0.4]

14. Secondary Outcome: Number of Participants With Adverse Events/Complications
Description: Comparing individual non-endpoint adverse events between ablative and drug therapy is difficult due to the substantial difference in the types of adverse events expected.
  Ablation-related events were counted among all patients that were randomized to and received an ablation.
  Drug-related events were counted among all patients that were randomized to and received drug therapy.
Time Frame: From treatment start date to date of event over a median follow-up of 48.5 months.
Population: Ablation-related events were counted among all patients that were randomized to and received an ablation.
  Drug-related events were counted among all patients that were randomized to and received drug therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
Number analyzed (Participants) | 1006 | 1092
Participants
  Hyper- or hyopthyroidism | 0 | 17
  Hypotension | 0 | 3
  Major proarrhythmic event (VT, VF) | 0 | 9
  Atrial proarrhythmic event | 0 | 1
  Allergic reaction | 0 | 7
  Gastrointestinal abnormality (excluding >moderate) | 0 | 3
  Liver injury/failure | 0 | 3
  Pulmonary toxicity | 0 | 1
  Hematoma | 23 | 0
  Pseudo aneurysm | 11 | 0
  Atrial venous fistula | 4 | 0
  Pneumothorax | 1 | 0
  Sepsis | 1 | 0
  Cardiac tamponade with perforation | 8 | 0
  Transient ischemic attack (TIA) | 3 | 0
  Myocardial infarction | 1 | 0
  Severe pericardial chest pain | 11 | 0
  Phrenic nerve injury | 1 | 0
  Pulmonary vein stenosis >75% | 1 | 0
  Esophageal ulcer | 5 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment through study completion over a median follow-up duration of 48.5 months.
Arm/Group | Left Atrial Ablation | Rate or Rhythm Control Therapy
All-Cause Mortality (participants affected / at risk) | 58/1108 | 67/1096
Serious Adverse Events (participants affected / at risk) | 454/1108 | 430/1096
Other Adverse Events (participants affected / at risk) | 0/1108 | 0/1096
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Left Atrial Ablation (N=1108) | Rate or Rhythm Control Therapy (N=1096)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
ANAEMIA OF MALIGNANT DISEASE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
AUTOIMMUNE HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HAEMORRHAGIC DISORDER (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IMMUNE THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (2) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 2 (2)
ANGINA PECTORIS (Cardiac disorders) | 7 (7) | 5 (5)
ANGINA UNSTABLE (Cardiac disorders) | 4 (4) | 4 (5)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 0 (0) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 7 (7) | 5 (6)
ATRIAL SEPTAL DEFECT ACQUIRED (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL TACHYCARDIA (Cardiac disorders) | 6 (8) | 1 (2)
ATRIAL THROMBOSIS (Cardiac disorders) | 2 (2) | 0 (0)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 7 (7) | 3 (3)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 18 (18) | 25 (28)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 10 (10) | 9 (10)
CARDIAC FAILURE (Cardiac disorders) | 60 (90) | 47 (77)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 4 (4) | 3 (3)
CARDIAC PERFORATION (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 10 (10) | 1 (1)
CARDIAC VALVE DISEASE (Cardiac disorders) | 4 (4) | 5 (5)
CARDIAC VENTRICULAR THROMBOSIS (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 9 (9) | 3 (3)
CORONARY ARTERY EMBOLISM (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 4 (5) | 6 (7)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 3 (3) | 1 (1)
INTRACARDIAC THROMBUS (Cardiac disorders) | 5 (5) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 2 (2)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 1 (1)
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 7 (8) | 18 (20)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 22 (24) | 3 (3)
PERICARDITIS (Cardiac disorders) | 8 (8) | 2 (2)
PERICARDITIS CONSTRICTIVE (Cardiac disorders) | 1 (1) | 0 (0)
SINOATRIAL BLOCK (Cardiac disorders) | 3 (3) | 4 (4)
SINUS ARREST (Cardiac disorders) | 1 (1) | 2 (2)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
SINUS NODE DYSFUNCTION (Cardiac disorders) | 10 (10) | 13 (13)
TACHYARRHYTHMIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
TACHYCARDIA INDUCED CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1)
TRICUSPID VALVE DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 2 (2)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 2 (2) | 3 (3)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 11 (13) | 9 (11)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
MUSCULAR DYSTROPHY (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
PATENT DUCTUS ARTERIOSUS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 (1) | 0 (0)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 0 (0) | 1 (1)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 (1) | 0 (0)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 0 (0) | 3 (3)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 3 (3)
CATARACT (Eye disorders) | 0 (0) | 2 (2)
CATARACT NUCLEAR (Eye disorders) | 0 (0) | 1 (1)
DIPLOPIA (Eye disorders) | 0 (0) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 0 (0) | 1 (1)
OPTIC NERVE DISORDER (Eye disorders) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 1 (1) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (2)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ALCOHOLIC PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 2 (2)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 2 (2)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (2)
DUODENAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC DISORDER (Gastrointestinal disorders) | 5 (5) | 4 (4)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 10 (10) | 10 (11)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 4 (4)
HAEMATEMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 3 (3)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (2)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 1 (2)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 4 (5)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 0 (0)
OESOPHAGEAL DISORDER (Gastrointestinal disorders) | 2 (2) | 1 (1)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 3 (3) | 0 (0)
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 (0) | 1 (1)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1)
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 2 (2)
RECTAL PROLAPSE (Gastrointestinal disorders) | 1 (2) | 0 (0)
RECTAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 3 (3)
SMALL INTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
SUBILEUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
TONGUE GEOGRAPHIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 4 (4)
VOMITING (Gastrointestinal disorders) | 6 (6) | 2 (2)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0)
CARDIAC DEATH (General disorders) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 4 (4) | 2 (2)
DEATH (General disorders) | 14 (14) | 11 (11)
DEVICE MALFUNCTION (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 2 (3) | 2 (2)
HERNIA (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 1 (1) | 0 (0)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (5) | 4 (4)
PAIN (General disorders) | 1 (1) | 4 (4)
PYREXIA (General disorders) | 1 (1) | 0 (0)
STENT-GRAFT ENDOLEAK (General disorders) | 0 (0) | 2 (2)
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 2 (2) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 5 (5) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 2 (2) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
CHRONIC HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 2 (2)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 3 (3)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1)
ABSCESS SOFT TISSUE (Infections and infestations) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
ANORECTAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (2) | 3 (3)
BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1)
BRONCHITIS (Infections and infestations) | 2 (2) | 1 (1)
CELLULITIS (Infections and infestations) | 7 (7) | 3 (3)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (2)
DIABETIC FOOT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIABETIC GANGRENE (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 3 (3) | 6 (7)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 2 (2) | 2 (2)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 1 (1)
INFECTION (Infections and infestations) | 11 (11) | 10 (11)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
LYME DISEASE (Infections and infestations) | 0 (0) | 2 (2)
MEDICAL DEVICE SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 32 (37) | 29 (34)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 3 (3) | 1 (1)
SALMONELLA BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 11 (12) | 11 (12)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STREPTOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 12 (12) | 10 (10)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
VULVAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BURN OESOPHAGEAL (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 7 (9) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
MENTAL STATUS CHANGES POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
NERVE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
POST CONCUSSION SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 11 (11) | 2 (3)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 11 (11) | 3 (3)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ANTICOAGULATION DRUG LEVEL ABOVE THERAPEUTIC (Investigations) | 0 (0) | 1 (1)
BLOOD BICARBONATE DECREASED (Investigations) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 3 (3)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 2 (2) | 1 (1)
INTERNATIONAL NORMALISED RATIO ABNORMAL (Investigations) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 10 (10) | 5 (5)
GOUT (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHONDROCALCINOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
GOUTY TOPHUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
MUSCLE DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 18 (21) | 24 (28)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
APPENDIX CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
CHOLANGIOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
DIFFUSE LARGE B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
INVASIVE LOBULAR BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARGE INTESTINE BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 4 (4)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PROSTATE CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF THE ORAL CAVITY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THROAT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY OCCLUSION (Nervous system disorders) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 2 (2)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 22 (22) | 33 (39)
CERVICAL MYELOPATHY (Nervous system disorders) | 0 (0) | 2 (2)
DEMENTIA (Nervous system disorders) | 1 (1) | 0 (0)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 7 (7) | 8 (8)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 3 (3) | 2 (2)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
HYPERTONIA (Nervous system disorders) | 1 (1) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
POST-INJECTION DELIRIUM SEDATION SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 2 (2)
RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 2 (2)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
SPINAL CORD HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 (3) | 2 (2)
SYNCOPE (Nervous system disorders) | 15 (17) | 19 (22)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 20 (20) | 19 (21)
TRIGEMINAL NEURITIS (Nervous system disorders) | 0 (0) | 1 (1)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 (0) | 1 (1)
VIITH NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0)
DEVICE BATTERY ISSUE (Product Issues) | 1 (1) | 0 (0)
DEVICE DAMAGE (Product Issues) | 0 (0) | 1 (1)
DEVICE DISLOCATION (Product Issues) | 1 (1) | 0 (0)
DEVICE INAPPROPRIATE SHOCK DELIVERY (Product Issues) | 1 (1) | 0 (0)
DEVICE ISSUE (Product Issues) | 1 (1) | 0 (0)
DEVICE OCCLUSION (Product Issues) | 0 (0) | 1 (1)
THROMBOSIS IN DEVICE (Product Issues) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 2 (2)
CALCULUS BLADDER (Renal and urinary disorders) | 1 (1) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 5 (5)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 3 (3)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 16 (18) | 9 (10)
RENAL HAEMORRHAGE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 3 (3)
RENAL MASS (Renal and urinary disorders) | 1 (1) | 0 (0)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL CYST (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 2 (4)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 3 (3) | 1 (1)
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 (0) | 2 (2)
OVARIAN MASS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 4 (6)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (12)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 9 (9)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
PULMONARY TOXICITY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PULMONARY VEIN STENOSIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (6)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
CYTOREDUCTIVE SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 0 (0) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1) | 0 (0)
IMPLANTABLE DEFIBRILLATOR REMOVAL (Surgical and medical procedures) | 0 (0) | 1 (1)
IMPLANTABLE DEFIBRILLATOR REPLACEMENT (Surgical and medical procedures) | 1 (1) | 0 (0)
AORTIC ANEURYSM (Vascular disorders) | 2 (2) | 1 (1)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 (0) | 1 (1)
AORTIC DILATATION (Vascular disorders) | 1 (1) | 0 (0)
AORTIC OCCLUSION (Vascular disorders) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 4 (4) | 1 (1)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 1 (1)
ARTERIOVENOUS FISTULA (Vascular disorders) | 2 (2) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 (2) | 1 (1)
EMBOLISM (Vascular disorders) | 2 (2) | 4 (4)
GRANULOMATOSIS WITH POLYANGIITIS (Vascular disorders) | 1 (1) | 0 (0)
HAEMATOMA (Vascular disorders) | 17 (17) | 3 (3)
HAEMORRHAGE (Vascular disorders) | 7 (9) | 9 (9)
HYPERTENSION (Vascular disorders) | 7 (8) | 10 (10)
HYPERTENSIVE CRISIS (Vascular disorders) | 9 (10) | 11 (14)
HYPOTENSION (Vascular disorders) | 8 (8) | 2 (2)
INTERMITTENT CLAUDICATION (Vascular disorders) | 1 (1) | 0 (0)
ISCHAEMIA (Vascular disorders) | 5 (6) | 10 (10)
LYMPHATIC FISTULA (Vascular disorders) | 1 (1) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL ARTERY THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 (1) | 1 (1)
VASCULAR STENOSIS (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study has been designed as a multicenter study and the data generated from Institution/PI's evaluation may not be sufficient to draw meaningful conclusions. Thus, Institution/PI shall not individually publish the results of the Study.

DOCUMENTS (2):
  • Study Protocol (2013-11-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT00911508/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT00911508/SAP_001.pdf